CLINICAL TRIAL: NCT06437405
Title: The Effects of a 12-Week Resistance Exercise Program Plus Vinegar Ingestion on Biomarkers of Intestinal Permeability, Cognition, and Mood State in Healthy Adults
Brief Title: Resistance Exercise Plus Vinegar Ingestion on Biomarkers in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Associate Dean, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00019774
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-05

CONDITIONS: LPS; Mood Disorders; Cognitive Change
Keywords: vinegar; resistance training; strength; depression
MeSH Terms: conditions — Mood Disorders; Depression | interventions — Acetic Acid

STUDY DESIGN:
Intervention Model Description: 12-week randomized controlled trial preceded by a 3-week control period
Who Masked: Participant
Masking Description: participants will be randomly assigned to the liquid vinegar group or the vinegar pill group (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liquid vinegar (Experimental): 2 tablespoons of liquid apple cider vinegar (5% acidity) diluted in one cup of water twice daily with meals providing 1.5g acetic acid.
  Interventions: Dietary Supplement: Vinegar liquid
- Vinegar pill (Placebo Comparator): one apple cider vinegar tablet (0.022g acetic acid) daily.
  Interventions: Dietary Supplement: vinegar pill

INTERVENTIONS:
Dietary Supplement: Vinegar liquid — one pill daily
  Other Names: Vinegar pill
  Arms: Liquid vinegar
Dietary Supplement: vinegar pill — One pill daily
  Arms: Vinegar pill

SUMMARY:
Given its capacity to stimulate exercise-induced neuroplasticity at lower doses compared to aerobic exercise, resistance exercise has become the top-recommended rehabilitation approach for individuals with neurocognitive impairments. Despite a large body of evidence supporting its application in the context of cognition, little work has been done to investigate the role of resistance exercise in modifying the structure and function of the microbiota-gut-brain axis. Likewise, despite a general understanding of the benefits of short chain fatty acids such as acetate for the gut-brain axis, the impact of exogenous acetic acid has not been sufficiently examined in the context of the intestinal barrier. While self-reported mood disturbance responds favorably to vinegar ingestion, it is currently unknown if these effects are also associated with changes in intestinal permeability.

DETAILED DESCRIPTION:
Existing resistance exercise interventions have produced promising outcomes indicating favorable shifts in microbial composition, intestinal barrier integrity, and serum biomarkers of inflammation. These changes appear to be particularly pronounced in individuals experiencing greater enhancements in lean mass, implying a crucial role for the hypertrophic effects of the exercise protocol. Given the current knowledge surrounding age-related cognitive decline and the pathophysiology of neurological and psychiatric disorders, it seems that many of the mechanisms significantly influenced by resistance exercise could contribute to reducing the risk or, at the very least, delaying the onset of these conditions. Considering the observed neuroplastic and neuroprotective effects of resistance exercise on the brain, it is plausible to hypothesize that the mitigation of excessive intestinal permeability and subsequent neuroinflammation may further support overall brain function. Given the potential for vinegar to enhance these outcomes, investigating the combined effects of exercise and vinegar ingestion may provide valuable insights into how lifestyle interventions can effectively promote cognitive and mental health. Therefore, the purpose of this work is to assess whether the combination of resistance exercise and vinegar ingestion elicits more favorable shifts in gut barrier function, cognition, and mental health compared to resistance exercise alone. This investigation aims to demonstrate the potential efficacy of this integrated approach in fostering long-team health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. premenopausal (for those assigned female at birth)
2. willing and able to participate in moderate to vigorous exercise as determined by the ACSM Health/Fitness Facility Preparticipation Screening Questionnaire
3. sedentary (defined as a score <14 on the Godin-Shepard Leisure Time Physical Activity Questionnaire (GSLTQ))
4. equipped with access to a complete gym
5. available for all lab visits (at weeks 0, 3, 9, and 15)

Exclusion Criteria:

1. antibiotic use within the past three months
2. prebiotic, probiotic, or high-dose antioxidant supplementation within the past month
3. regular engagement in moderate to vigorous exercise
4. following a vegetarian diet
5. presence of any medical/psychiatric disease
6. presence of any gastrointestinal disorder such as irritable bowel syndrome, inflammatory bowel disease, Crohn's disease, diverticulitis/diverticulosis, etc.
7. actively pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Lipopolysaccharide | 12 weeks
  measured indirectly via LPS binding protein
Depression | 12 weeks
  measured via Profile of Mood States (POMS) questionnaire
Cognitive change | 12 weeks
  measured using Trail Making Test

CONTACTS AND LOCATIONS:
Locations (1):
- 850 PBC, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data beyond study investigators.